CLINICAL TRIAL: NCT00801541
Title: Characterization of Early Markers of Choroidal Neovascularization in Fellow Eyes of Patients With AMD and CNV in One Eye. (CNV-Markers)
Brief Title: Characterization of Early Markers of Choroidal Neovascularization
Acronym: CNV-Markers
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: CNTM326_A9010002
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2014-04

CONDITIONS: Age-related Macular Degeneration
Keywords: AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AMD: Patients with wet AMD in one eye and dry AMD in the other eye (study eye).

SUMMARY:
To this study and identify the sequence of alterations occurring in the chorioretinal interface during progression of AMD from "dry" AMD to sight-threatening chorioretinal neovascularization (CNV).

DETAILED DESCRIPTION:
The primary statistical objective of this study is to identify the sequence of alterations occurring in the chorioretinal interface during progression of AMD from risk "dry" AMD to sight-threatening chorioretinal neovascularization (CNV) (wet AMD).

Different imaging methods will be used simultaneously and at regular intervals in order to characterize markers or predictors of conversion to sight-threatening CNV will be: CNV (classic or occult) or position of CNV within 2500 µm (~1.7 disc diameters) of the foveal center, as evidenced by fluorescein angiography.

This is an institutional, prospective, observation study to be performed in fellow eyes of patients with evidence of "wet" AMD in other eye. Therefore, patients will have evidence of exudative ("wet") AMD in one eye ( the non-study eye) and non-exudative ("dry") AMD in the fellow eye (the study eye) that is at risk for progressive to exudation "wet" CNV.

Patients will exit the study at the time of developing sight-threatening CNV in the study eye and will be treated at the discretion of the physician.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age over 50 years
* Any race and any sex
* Clinical diagnosis of exudative AM;D in one eye (non-stud eye) and the presence of the following characteristics in the second eye (study eye, eye to be treated):

  * At least 5 or more intermediate (> 63 µm) or larger soft drusen AND/OR Confluent drusen within 3000 µm of the fovea center
  * Hyperpigmentation

Exclusion Criteria:

* History of medical condition that would preclude scheduled study visits
* History of ophthalmic disease in the study eye other than AMD
* Clinical signs of myopic retinopathy, or refraction higher than -8 diopter power.
* Intraocular surgery in the study eye within 60 days prior enrollement
* Evidence of past or present CNV in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of either sex, any race, aged over 50 years and over, diagnosed with exudative (wet) AMD in one eye (non-study eye) and non-exudative (dry) AMD (intermediate or large/confluent drusen, with hyperpigmentation, and no CNV or geographic atrophy) in the other eye (study eye) that is at risk for progressing to exudative (wet) AMD and meet all the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Wet AMD development in the study eye. | Single Visit

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, MD PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI - Clinical Trial Center, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Derived] Marques JP, Costa M, Melo P, Oliveira CM, Pires I, Cachulo ML, Figueira J, Silva R. Ocular Risk Factors for Exudative AMD: A Novel Semiautomated Grading System. ISRN Ophthalmol. 2013 Jul 30;2013:464218. doi: 10.1155/2013/464218. eCollection 2013. PMID 24555130
- See also: Related Info — http://www.aibili.pt